CLINICAL TRIAL: NCT04775706
Title: A Multicenter, Proof-of-concept, Phase 2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HM15912 (Sonefpeglutide) in Adult Subjects With Short Bowel Syndrome-associated Intestinal Failure (SBS-IF)
Brief Title: Phase 2 Study to Assess the Safety, PK, and PD of Sonefpeglutide (HM15912) in SBS-IF Subjects
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-GLP2-201; DOLPHINS-2 (Other: Hanmi Pharm. Co., Ltd.)
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-03

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HM15912 0.5 mg/kg, 1.0mg/kg, 1.5mg/kg Active (Experimental)
  Interventions: Drug: HM15912 Active
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HM15912 Active — Randomized, double-blind, placebo-controlled
  Arms: HM15912 0.5 mg/kg, 1.0mg/kg, 1.5mg/kg Active
Drug: Placebo — Randomized, double-blind, placebo-controlled
  Arms: Matching Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, proof-of-concept (PoC), Phase 2 study to assess the safety, PK, and PD of SC administration of HM15912(sonefpeglutide) in adult subjects with SBS-associated intestinal failure (SBS-IF).

DETAILED DESCRIPTION:
The study consists of a screening period, a run-in period, a 6-months core treatment period, a 7-months extension treatment period and a 1-month safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, aged 18 years of age or older with SBS resulting in intestinal failure at the time of signing the informed consent form (ICF) (or country's legal age of majority if the legal age is <18 years)
2. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol
3. Diagnosis of SBS with the latest intestinal resection being at least 6 months prior to Screening and considered stable regarding the PN/IV need. No restorative surgery planned in the study period.

Exclusion Criteria:

1. Any history of colon cancer.
2. History of any other cancers (except margin-free resected cutaneous basal or squamous cell carcinoma or adequately treated in situ cervical cancer) unless disease-free for at least 5 years
3. History of alcohol or drug abuse (within 1 year of screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | for 24 weeks
  after multiple subcutaneous (SC) doses

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - The Cleveland Clinic Foundation, Cleveland, Ohio
- UZ Leuven, Leuven, Vlaams Brabant, Belgium
- Rigshospitalet Department of Digestive Diseases, Transplantation and General Surgery Section for Intestinal Failure, Copenhagen, Denmark
- France (4):
  - Hopital Beaujon, Clichy, Clichy
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Les Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Universitaire de Nice, Nice
- Germany (2):
  - Asklepios Klinik St. Georg, Hamburg, Hamburg
  - Universitätsklinikum Tübingen, Tübingen, Tübingen
- Wojewodzki Specjalistyczny Szpital im. Mikołaja Pirogowa w Łodzi, Lodz, Łódź Voivodeship, Poland
- Samsung Medical Center, Seoul, South Korea
- Central Middlesex Hospital, London, United Kingdom